CLINICAL TRIAL: NCT01948713
Title: Effect of Pelvic Floor and Hip Muscle Strengthening in the Treatment of Stress Urinary Incontinence: Randomized Blind Clinical Trial
Brief Title: Effect of Pelvic Floor and Hip Muscle Strengthening in the Treatment of Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SimoneM
Record Dates: First submitted 2013-06-05; First posted 2013-09-24 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Strengthening of pelvic floor muscles.
  Interventions: Other: Strengthening of pelvic floor muscles.
- Group 2 (Experimental): Strengthening of pelvic floor muscles associated with strengthening of hip muscles.
  Interventions: Other: Strengthening of pelvic floor muscles.; Other: Strengthening of hip muscles.

INTERVENTIONS:
Other: Strengthening of pelvic floor muscles. — Kegel exercises kinesiotherapy
Other: Strengthening of hip muscles. — Kegel exercises and strengthening of hip muscles as Gluteus Maximus and Medius and adductor muscles
  Arms: Group 2

SUMMARY:
INTRODUCTION: Stress urinary incontinence is a common condition in women and can be defined as the involuntary loss of urine on exertion, exercise, sneezing or coughing. This pathology causes physical discomfort and impacts the quality of life in a negative manner. Physiotherapeutic exercises is a treatment with low cost and high patient attendance. It can be applied with focus on strengthening the pelvic floor muscles or on muscular synergism. OBJECTIVE: To compare the effectiveness of Kegel exercises performed alone or performed in association with the strengthening of the muscles of the hip in the treatment of stress urinary incontinence. METHODOLOGY: The study is a randomized, blinded clinical trial. It aims at assessing objectively the strength of the pelvic floor, the improvement in the number of episodes of loss and impact on quality of life. The study will accept up to 40 women, who will be divided into two groups of physical therapy: group 1 (that will strengthen the pelvic floor muscles with Kegel exercises) and group 2 (that will perform strengthening the pelvic floor muscles with Kegel exercises associated with the strengthening of muscles of the hip). The two groups will be evaluated at the beginning and at the end of treatment.

DETAILED DESCRIPTION:
the strength of the pelvic floor muscles will be evaluated with the aid of a perineometer

ELIGIBILITY:
Inclusion Criteria:

* Women with 30 to 70 years of age;
* Clinical diagnosis of stress urinary incontinence;
* Urodynamic study.

Exclusion Criteria:

* Stress urinary incontinence with sphincter deficiency;
* Urinary urgence;
* Mixed urinary incontinence;
* Pregnant women;
* Neurological or muscular disease that interfere with continence;
* Urinary infection;
* Genital prolapse;
* Gynecological surgery for urinary incontinence in the last year;
* Hormone replacement therapy;
* Strength 0 in functional evaluation of the pelvic floor muscles.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-01-07 (Actual); Primary Completion 2014-09-18 (Actual); Study Completion 2015-01-08 (Actual)

PRIMARY OUTCOMES:
Change in frequence of urinary incontinence | At the first session of physical therapy and after 10 weeks of physical therapy treatment a voiding diary will be applied, and every session a follow up diary will be used. The physiotherapy treatment will be held twice a week for 10 weeks.
  number of episodes of urinary leakage per week

SECONDARY OUTCOMES:
Change in strength of pelvic floor muscles | At the first session of physical therapy and after 10 weeks of physical therapy treatment . The physiotherapy treatment will be held twice a week for 10 weeks.
  The strength of pelvic floor muscles will be assessed qualitatively by the functional evaluation of pelvic floor and quantitatively by perineometer.
Change in quality of life | At the first session of physical therapy and after 10 weeks of physical therapy treatment . The physiotherapy treatment will be held twice a week for 10 weeks.
  Questionnaires: International Consultation on Incontinence Questionnaire (ICIQ); King´s Health Questionnaire (KHQ)

CONTACTS AND LOCATIONS:
Overall Officials: Simone A. Marques, researcher, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322